## Statistical Analysis Plan (SAP)

For Protocol: USUHS-20250225

Last Updated: June 5, 2025

## 1.0 Outcome Measures

- Co-primary Outcome Measures:
  - Comparison between TBI and AHI groups in the percent change in migraine headache
    - **frequency** from baseline to peak effect.
  - Comparison between TBI and AHI groups in the percent change in migraine headache
    - intensity from baseline to peak effect.
  - Comparison between TBI and AHI groups in the percent change in HIT-6 score from baseline to peak effect.
- Secondary Outcome Measures: Secondary outcomes include comparing absolute changes in frequency, intensity, and HIT-6 scores; changes in other migraine characteristics; timelines of Xeomin effectiveness; and assessment of residual effects after the treatment has worn off.

## 2.0 Sample Size and Power

- Sample Size: The estimated sample size is 40 patients in the TBI group and 20 patients in the AHI group. This is a convenience sample based on clinic availability.
- Statistical Power: With a two-sided alpha of 0.05, the study has a power of 0.8 to detect Cohen's d effect sizes of 0.799 using Mann-Whitney U tests, which is considered a moderate to large effect size.

## 3.0 Data Analysis Plan

 Assumptions: The analysis assumes that the data distributions for the TBI and AHI groups will not be normal; therefore, non-parametric statistical methods will be used.

- Quantitative Variables: Medians and 25-75%iles will be calculated. Two-sided Mann-Whitney U tests will be used to compare quantitative variables between the TBI and AHI groups, with Cohen's d calculated to measure effect size.
- Qualitative Variables: Frequencies and percentages will be calculated.
  Chi-squared tests will be used for comparisons between the TBI and AHI groups.
- Missing Data and Outliers:
  - Missing Data: Missing primary outcome data will be handled with case-wise deletion. Missing secondary outcome data will be imputed using multivariable interpolation, with sensitivity analyses conducted.
  - Outliers: Outliers will be examined, and if deemed genuine, they will be retained and noted in the results, as they may be of clinical interest. The non-parametric methods are expected to be robust to outliers.
- **Subgroup Analyses:** Exploratory subgroup analyses based on factors like age, sex, and migraine history may be conducted.
- **Interpretation:** Given this is the first study of its kind, results will require replication and statistical correction for multiple comparisons will not be performed.